CLINICAL TRIAL: NCT00349011
Title: Menopausal Therapy in Women at Increased Risk for Breast Cancer: Does a Personalized Risk Assessment and Counseling Intervention Aid in Decision-Making?
Brief Title: Genetic Counseling for Menopausal Therapy Decision-Making for Women at Increased Risk for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Massachusetts General Hospital (Other); Women and Infants Hospital of Rhode Island (Other); Stony Brook University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: Komen BCTR0100202
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Menopause
Keywords: menopause; genetic counseling; breast cancer; tamoxifen; chemoprevention
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: Personalized risk assessment
Procedure: genetic counseling intervention

SUMMARY:
The purpose of this study is to determine the effects of a personalized menopausal therapy risk assessment and genetic counseling intervention on knowledge, risk perception, and decision-making in healthy women at increased risk for breast cancer.

DETAILED DESCRIPTION:
Women with a family history of breast cancer have several menopausal therapy options, including tamoxifen, hormone therapy, alternative medications, or no treatment. This complex decision should be based on each woman's risk to develop breast cancer, menopausal symptoms, preferences, and risks for other conditions. Current models in use for menopausal therapy counseling do not include pedigree analysis, personalized risk assessment or genetic testing in this process. The purpose of this multi-center study is to determine the effects of a personalized risk assessment and genetic counseling intervention on knowledge, risk perception, and decision-making in a group of healthy women who had a first-degree relative with breast cancer. Intervention participants will be given a personalized risk assessment for breast cancer, heart disease, osteoporosis, and uterine cancer based on family history and personal health data.

ELIGIBILITY:
Inclusion Criteria:

* at least one first degree relative with breast cancer
* age 40 or older

Exclusion Criteria:

* currently taking a menopausal therapy
* previous cancer diagnosis (except basal cell carcinoma)
* previous diagnosis of atypical hyperplasia
* previous diagnosis of lobular carcinoma in situ (LCIS)
* known carrier of a BRCA1 or BRCA2 mutation
* personal history of heart disease
* >10% risk of carrying a BRCA1 or BRCA2 mutation

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-08; Study Completion 2004-03

PRIMARY OUTCOMES:
Decisional conflict
Knowledge of menopause and menopausal therapy
Satisfaction with counseling intervention
Medication usage

SECONDARY OUTCOMES:
Perceived risk of breast cancer, heart disease, osteoporosis
Worry about breast cancer, heart disease, osteoporosis

CONTACTS AND LOCATIONS:
Overall Officials: Ellen T. Matloff, M.S., Principal Investigator — Yale University
Locations (1):
- Yale Cancer Genetic Counseling, Yale Cancer Center, Yale University School of Medicine, New Haven, Connecticut, United States